CLINICAL TRIAL: NCT01291095
Title: Phase II Randomized Controlled Trial of Accelerated Fractionation Radiotherapy (6 Fractions Per Week) Versus Concurrent Chemoradiotherapy in Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Accelerated Fractionation Radiotherapy (AFRT) Versus Concurrent Chemoradiotherapy (Crt) In Locally Advanced Head And Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: DR SUDEEP DAS, ALL INDIA INSTITUTE OF MEDICAL SCIENCES, NEW DELHI, INDIA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCTOFAFRTVSCRTINHNSCCAIIMS
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: HEAD AND NECK CANCER
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CONCURRENT CHEMO-RADIOTHERAPY ARM (Active Comparator): Patients assigned to CRT arm will be given radiation one fraction per day, on five consecutive days from Monday to Friday along with intravenous cisplatin 40 mg/m2 weekly for seven doses (a minimum of 5weekly chemotherapy).
  Interventions: Drug: CISPLATIN; Radiation: EXTERNAL BEAM RADIOTHERAPY
- ACCELERATED FRACTIONATION RADIOTHERAPY ARM (Experimental): Patients assigned to AFRT arm will undergo radiation similarly one fraction per day and then the sixth fraction will be given on another day (Saturday) or as an extra fraction on one of the first five days, but always allowing at least a 6-hour interval between fractions on same day. If any unintended interruption of the treatment occurs, this missing treatment will be given as soon as possible, preferably within a week, but not allowing more than 14 Gy to be given during any 7-day period.
  Interventions: Radiation: EXTERNAL BEAM RADIOTHERAPY

INTERVENTIONS:
Drug: CISPLATIN — IN CRT ARM:RADIATION ONE FRACTION PER DAY, ON FIVE CONSECUTIVE DAYS FROM MONDAY TO FRIDAY ALONG WITH INTRAVENOUS CISPLATIN 40mg/m2 WEEKLY FOR SEVEN DOSES.
  IN AFRT ARM: PATIENTS WILL NOT RECEIVE ANY CHEMOTHERAPY WITH CISPLATIN
  Other Names: CDDP
  Arms: CONCURRENT CHEMO-RADIOTHERAPY ARM
Radiation: EXTERNAL BEAM RADIOTHERAPY — Patients assigned to CRT arm will be given radiation one fraction per day, on five consecutive days from Monday to Friday along with intravenous cisplatin 40 mg/m2 weekly for seven doses (a minimum of 5weekly chemotherapy). Patients assigned to AFRT arm will undergo radiation similarly one fraction per day and then the sixth fraction will be given on another day (Saturday) or as an extra fraction on one of the first five days, but always allowing at least a 6-hour interval between fractions on same day. If any unintended interruption of the treatment occurs, this missing treatment will be given as soon as possible, preferably within a week, but not allowing more than 14 Gy to be given during any 7-day period.
  Other Names: EBRT

SUMMARY:
The aim of this trial is to compare the accelerated fractionation radiotherapy and concurrent chemo-radiotherapy in locally advanced head and neck squamous cell carcinoma patients in terms of loco-regional control, toxicities and quality of life.

DETAILED DESCRIPTION:
Concurrent chemo-radiotherapy is a common and conventional method of treating locally advanced head and neck squamous cell carcinoma (HNSCC). In locally advanced HNSCC it has been proved to be superior to radiotherapy alone. On the other side accelerated fractionation radiotherapy (AFRT) is a proven practice to improve cure rate in head and neck cancers. Yet it has not been compared with Concurrent Chemoradiotherapy (CRT) in locally advanced HNSCC and hence this study is aiming to compare CRT versus AFRT.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20 - 60 years old
2. Karnofsky performance scale score 70 or above
3. Biopsy proven squamous cell carcinomas (SCC) of oropharynx, larynx and hypopharynx
4. TNM stages- Stage III -IVB
5. Informed consent (in prescribed form under institutional guidelines)

Exclusion Criteria:

1. Lack of histopathological proof of malignancy (HNSCC)
2. Doubtful follow-up and/ or non-compliance
3. Previous oncologic therapy with surgery, radiotherapy or chemotherapy
4. Uncontrolled comorbid conditions e.g hypertension, diabetes mellitus, chronic obstructive pulmonary disease, coronary artery disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
TO COMPARE THE LOCO-REGIONAL TUMOR CONTROL RATE BETWEEN AFRT & CRT IN LOCALLY ADVANCED HEAD AND NECK SQUAMOUS CELL CARCINOMAS. | 5months(2months treatment period followed by 3 months observation)
  To compare the loco-regional tumor control rate clinical assessment after 3months of treatment completion will be done.CECT of face and neck at 3 months post treatment completion will be done.
TO COMPARE THE TOXICITY BETWEEN AFRT AND CRT IN LOCALLY ADVANCED HEAD AND NECK SQUAMOUS CELL CARCINOMAS | 3 months(2 month treatment periods followed by 1month observation)
  To compare toxicity weekly and at 1month post treatment completion hemogram will be done and assessed by CTCAE V3.0. Assessment of acute morbidity clinically will be done by CTCAE V-3.0 scoring system weekly, and post-RT 1 month.

SECONDARY OUTCOMES:
TO COMPARE POST-THERAPY QUALITY OF LIFE BETWEEN AFRT AND CRT IN LOCALLY ADVANCED HEAD AND NECK SQUAMOUS CELL CARCINOMA. | 5months(2months treatment period followed by 3months observation)
  TO COMPARE THE POST-THERAPY QUALITY OF LIFE BETWEEN AFRT AND CRT IN LOCALLY ADVANCED HNSCC.Assessment of quality of life in patients in both arms will be recorded prior to start of treatment(for base-line record) and subsequently at 1month and 3months after treatment completion using European organization for research and treatment in cancer, Belgium quality of life questionnaire (EORTC QLQ-C30 & QLQ-H&N35).

CONTACTS AND LOCATIONS:
Overall Officials: Dr SUDEEP DAS, MBBS, Principal Investigator — ALL INDIA INSTITUTE OF MEDICAL SCIENCES, NEW DELHI, INDIA
Locations (1):
- Dr B.R.A.I.R.C.H, ALL INDIA INSTITUTE OF MEDICAL SCIENCES, NEW DELHI, New Delhi, Other State, India